CLINICAL TRIAL: NCT00859911
Title: The Effectiveness of Multiple Micronutrient Supplements Given by Teachers to School-Age Children on Growth and Educational Achievement
Brief Title: The Effectiveness of Micronutrient Supplements on Growth and Educational Achievement of Schoolchildren in Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Save the Children (Other)
Collaborators: University of Westminster (Other); Harvard University (Other)
Responsible Party: Andrew Hall, University of Westminster
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCBD01
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Micronutrient Deficiencies
Keywords: micronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Thiamine Mononitrate 5mg, Riboflavin 2 mg, Niacin amide 20 mg, Pyridoxine hydrochloride 2 mg
  Interventions: Dietary Supplement: Multiple micronutrients
- 1 (Experimental): Vitamin A 1500 µg, Vitamin D 15 µg, Thiamine Mononitrate 1.22 mg, Riboflavin 1.7 mg, Ascorbic Acid 60 mg, Niacin amide 20 mg, Pyridoxine hydrochloride 2 mg, Folic Acid 400 µg, Calcium pantothenate 10.8 mg, Cyanocobalamin 6 µg, Vitamin E 18 IU, ferrous sulphate 19 mg, potassium iodide 145 µg, Potassium sulphate 11 mg, Manganese sulphate 0.38 mg, copper sulphate 0.509 mg, zinc sulphate 15 mg
  Interventions: Dietary Supplement: Multiple micronutrients

INTERVENTIONS:
Dietary Supplement: Multiple micronutrients — A tablet on three days a week containing: Vitamin A 1500 µg, Vitamin D 15 µg, Thiamine Mononitrate 1.22 mg, Riboflavin 1.7 mg, Ascorbic Acid 60 mg, Niacin amide 20 mg, Pyridoxine hydrochloride 2 mg, Folic Acid 400 µg, Calcium pantothenate 10.8 mg, Cyanocoblamin 6 µg, Vitamin E 18 IU, ferrous sulphate 19 mg, potassium iodide 145 µg, Potassium sulphate 11 mg, Manganese sulphate 0.38 mg, copper sulphate 0.509 mg, zinc sulphate 15 mg
  Other Names: V-Plex Plus, Acme Pharmaceuticals Bangladesh

SUMMARY:
This is a study of the effectiveness of multiple micronutrient supplements given by teachers to their pupils on growth and educational achievements. The hypothesis is that children are deficient in multiple micronutrients and that supplements will lead to improved weight gain, growth in height and better educational achievements in tests of mathematics and language. It is also hypothesised that micronutrients will help prevent the build up of arsenic consumed in food and water as a result of geological contamination of water sources.

DETAILED DESCRIPTION:
This study is a randomised double blind controlled cluster trial of the effectiveness of multiple micronutrient supplements given by teachers to schoolchildren on improving their growth, nutritional status and educational achievement. The primary outcome measures are: gains in weight and height, haemoglobin concentration, cognitive function and educational achievement. Secondary outcomes are other anthropometric measurements and a decrease in body arsenic deposits. One hundred schools in Meherpur District, Bangladesh will take part in this study. Participation will be on the basis of informed consent. All pupils will be dewormed twice a year using a single dose of 400 mg albendazole; this will promote the bioavailability of the micronutrient supplements. The schools will be randomly allocated into two groups. In one group of 50 schools all children will be given by their teachers a single tablet of multiple micronutrients on every other school day each week, so for a total of 3 days a week or about 125 school days a year, depending on school and national holidays. This supplement will make a substantial contribution over a period of one year to each child's recommended intake of iron, iodine, zinc, vitamin A, vitamin B12, folate and four B-group vitamins. Some of these micronutrients, such as vitamin A and iron, can be stored in the body, in addition to meeting current nutritional requirements. Children in the other 50 schools will receive a tablet identical in weight, shape, size and appearance that contains the same four B-group vitamins as the multiple micronutrient supplement. The B-group vitamins are not expected to have a major effect on any of the outcome measures, but may provide some benefit to children in the comparison group. Both supplements are formulated according to UK and US pharmacopoeias by Acme Pharmaceuticals and are being purchased by Save the Children. Both supplements will be given free on three days a week to an estimated 30,000 pupils in all 100 study schools for a period of two school years. The subjects for study will be up to 30 randomly selected children in class 2 in the age range 7 - 8 years in all 100 schools. An equal number of boys and girls will be selected. The actual number will depend on enrolment in class 2 in each school. A baseline survey will be done before the supplements are started to measure the following: weight, height and other anthropometric measurements to assess growth; the prevalence of intestinal worm infections in a 20% sub-sample; the haemoglobin concentration in a drop of blood taken from a finger prick from a sub-sample of about 66% of all children; the concentration of arsenic in hair in a sub-sample of about 20% of all children; tests of cognitive function including concentration in all children; and tests of educational achievement in mathematics and language in all children. These measurements, analyses and assessments will be repeated two years later when the cohort of up to 1,500 children in each study group are in class 4. The magnitude and statistical significance of differences in the mean differences in outcome values between study groups will indicate the impact of the multiple micronutrient supplement in comparison with B-group vitamins alone.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in class 2
* Parents and child consented

Exclusion Criteria:

* Severely anaemic
* Physically disabled

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
tests of educational achievement and concentration | 2 years
gains in weight and height | 2 years

SECONDARY OUTCOMES:
haemoglobin concentration | 2 years
concentration of arsenic in hair | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hall, PhD, Principal Investigator — University of Westminster
Locations (1):
- Save the Children, Dhaka, Dhaka Division, Bangladesh